CLINICAL TRIAL: NCT02073721
Title: The Importance of Electrical Stimulation as a Treatment for Urinary Incontinence in Patients Undergoing Prostatectomy to Exercise the Pelvic Floor Muscles (MAPs): Randomised Controlled Trial, Double Blind
Brief Title: The Importance of Electrical Stimulation as a Treatment for Urinary Incontinence in Patients Prostatectomy
Acronym: UI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Gama Filho (Other)
Responsible Party: Principal Investigator, Patrícia Zaidan de Barros, Electrostimulation exercises of the pelvic floor muscles AND URINARY INCONTINENCE IN POST prostatectomy: Randomised controlled trial, double blind, Universidade Gama Filho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 260535
Record Dates: First submitted 2013-06-01; First posted 2014-02-27 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- electrostimulation with exercises MAPs (Experimental): this group will make the electrostimulation with exercises of the pelvic floor muscles with a focus on strengthening the pelvic floor muscles.
  Interventions: Other: electrostimulation with exercises MAPs
- exercises MAPs (Active Comparator): This group will focus exercises of the pelvic floor muscles with strengthening the muscles of the pelvic floor
  Interventions: Other: exercises MAPs

INTERVENTIONS:
Other: electrostimulation with exercises MAPs — this group will make the electrostimulation with exercises of the pelvic floor muscles with a focus on strengthening the pelvic floor muscles.the frequency will be 20 sessions, 2 times per week, lasting 30 minutes.
  Other Names: electrostimulation and exercises of the pelvic floor muscles
  Arms: electrostimulation with exercises MAPs
Other: exercises MAPs — This group will focus exercises of the pelvic floor muscles with strengthening the muscles of the pelvic floor. the frequency will be 20 sessions, 2 times per week, lasting 30 minutes.
  Other Names: exercises of the pelvic floor muscles
  Arms: exercises MAPs

SUMMARY:
The use of electrical stimulation to reduce urinary incontinence in men undergoing prostatectomy exercises of the pelvic floor muscles (MAPs)

DETAILED DESCRIPTION:
The study will be an experiment with active control, randomized, double-blind, parallel intervention. After met the eligibility criteria of the patients will be randomly allocated into two groups: Group exercises MAPs (GEX), which is the active control group and electrostimulation + exercises MAPs (GEEX).

ELIGIBILITY:
Inclusion Criteria:

* patients with urinary sphincter deficiency resulting from a radical prostatectomy surgery
* sent by urologists the same hospital where the experiment will take place
* having the maximum time six months after surgery
* to use 2 to 5 disposable protective per day

Exclusion Criteria:

* Symptoms of urinary tract infection
* symptoms of lower urinary tract obstruction
* anal fistula
* metallic implant in the body
* transurethral resection of prostate
* radiation therapy
* non-enforcement of the proposed treatment.

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
urinary incontinence | august/2013 to December/2013 (4 months)

CONTACTS AND LOCATIONS:
Overall Officials: Patrícia Z Barros, expert, Principal Investigator — Gama Filho University
Locations (1):
- Federal Hospital Servants of the State of Rio de Janeiro, Rio de Janeiro, RJ/Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Johnson EE, Mamoulakis C, Stoniute A, Omar MI, Sinha S. Conservative interventions for managing urinary incontinence after prostate surgery. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD014799. doi: 10.1002/14651858.CD014799.pub2. PMID 37070660